CLINICAL TRIAL: NCT01998724
Title: Tai Chi After Pulmonary Rehabilitation in Patients With COPD: A Randomized Trial
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012P000220; R01AT006358 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic bronchitis; Emphysema; Pulmonary; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (No Intervention): No intervention
- Tai Chi Exercise (Experimental): 24 week Tai Chi intervention designed for individuals with COPD
  Interventions: Behavioral: Tai Chi
- Group Walking Exercise (Experimental): 24 week group walking intervention
  Interventions: Behavioral: Group Walking

INTERVENTIONS:
Behavioral: Tai Chi — 24 week tai chi intervention designed for individuals with COPD
  Arms: Tai Chi Exercise
Behavioral: Group Walking — 24 week group walking intervention
  Arms: Group Walking Exercise

SUMMARY:
The main purpose of this study is to determine the feasibility and effects of a 6-month tai chi exercise program as compared to a 6-month group walking program and standard care for patients with COPD that have recently completed a pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

1. COPD defined as FEV1 (Forced expiratory volume in 1 second)/FVC (Forced vital capacity) <0.70 or chest CT evidence of emphysema
2. Age > 40 years
3. Any severity of COPD as defined by GOLD (Global Obstructive Lung Disease) stages 1, 2,3, or 4
4. Completion of standard pulmonary rehabilitation of at least 8 weeks duration within 24 weeks prior to study entry* *Defined as attending 65% of the program's sessions with a minimum of 10 sessions

Exclusion Criteria:

1. COPD exacerbation requiring steroids, antibiotics, ED visit or hospitalization within the past 2 weeks unless physician deems subject at baseline
2. Hypoxemia on walk test (O2 sat < 85% on oxygen)
3. Inability to ambulate due to vascular or other neuromuscular conditions that would preclude a walk test
4. Clinical signs of unstable cardiovascular disease (ie. chest pain on walk test)
5. Severe cognitive dysfunction (documented Mini-Mental Status Exam ≤ 24)
6. Non-English speaking
7. Current regular practice of tai chi
8. Current diagnosis of lung cancer or treated for lung cancer within the past 5 years
9. Unstable/untreated mental health issue that precludes informed consent or otherwise affects ability to participate in the intervention

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of tai chi intervention | 24 weeks
  Willingness to participate, adherence, and safety

SECONDARY OUTCOMES:
Change from baseline - Disease specific quality of life | Baseline, 12 weeks, 24 weeks, 1 year
  Chronic Respiratory Questionnaire
Change from baseline - Exercise capacity | Baseline, 12 weeks, 24 weeks
  Six minute walk distance
Change from baseline - Dyspnea | Baseline, 12 weeks, 24 weeks, 1 year
  University of California, San Diego Shortness of Breath Questionnaire
Change from baseline - Psychosocial well-being | Baseline, 12 weeks, 24 weeks, 1 year
  Center for Epidemiologic Studies Depression Scale, Perceived Stress Scale, COPD Self-Efficacy Scale, Multidimensional Scale of Perceived Social Support
Changes from baseline - Pulmonary function | Baseline, 12 weeks, 24 weeks
  Spirometry
Change from baseline - Exercise Efficacy | Throughout study
  Daily exercise activities, step counts taken at baseline, 12 weeks, 24 weeks, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Yeh, MD, MPH, Principal Investigator — BIDMC, Harvard Medical School
Locations (2):
- United States (2):
  - VA Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Gilliam EA, Kilgore KL, Liu Y, Bernier L, Criscitiello S, Litrownik D, Wayne PM, Moy ML, Yeh GY. Managing the experience of breathlessness with Tai Chi: A qualitative analysis from a randomized controlled trial in COPD. Respir Med. 2021 Aug;184:106463. doi: 10.1016/j.rmed.2021.106463. Epub 2021 May 15. PMID 34023739
- [Derived] Moy ML, Wayne PM, Litrownik D, Beach D, Klings ES, Davis RB, Yeh GY. Long-term Exercise After Pulmonary Rehabilitation (LEAP): Design and rationale of a randomized controlled trial of Tai Chi. Contemp Clin Trials. 2015 Nov;45(Pt B):458-467. doi: 10.1016/j.cct.2015.09.004. Epub 2015 Sep 8. PMID 26362690